CLINICAL TRIAL: NCT03164343
Title: Pain Neuroscience Education in Healthy Children: A Pilot Study
Brief Title: Pain Neuroscience Education in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Roselien Pas, Principal investigator, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eduvalid Study (Part 2)
Record Dates: First submitted 2017-05-17; First posted 2017-05-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Child; Pain
Keywords: Pain Neuroscience Education
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Neuroscience Education for children (Experimental): All participants within this study will receive Pain Neuroscience Education
  Interventions: Device: Pain Neuroscience Education for children

INTERVENTIONS:
Device: Pain Neuroscience Education for children — Children and their parent will receive a +/- 1h one-on-one educational session about the neurophysiology of pain, adjusted to the child's comprehension status. Parents will be present in the PNE session too. The PNE program for children contains two sections: (1) The healthy pain system and its function, divided in subsections each consisting of a specific neurophysiological pain concept (i.e. central nervous system anatomy, nociception and nociceptive pathways, up- and down-regulation of the nervous system) and (2) adaptations of the pain system following persistent pain. To ensure interaction between therapist and child, an interactive board game was developed and used throughout the full educational session.

SUMMARY:
The primary objective of this study is to examine whether Pain Neuroscience Education for children is able to increase a child's knowledge on the neurophysiology of pain.

In addition, this study investigates the influence of PNE on several pain related outcomes; pain-related fear, pain catastrophizing and pain vigilance and awareness.

DETAILED DESCRIPTION:
Pain is a common and daily experience among children that is usually short-term, causing little to moderate discomfort. Yet, a substantial number of children experience chronic pain. Persistent pain periods mainly affect the children's school attendance and participation in recreational activities, possibly leading to academic impairments and social exclusion. Even worse is the children's greater predisposition to develop chronic pain into adulthood. Considering these disadvantages, children suffering from chronic pain should be treated as fast as possible and in the most optimal way. The existing literature on management in children with chronic pain encourages a multidisciplinary approach involving physical therapy and psychological interventions (i.e. cognitive behavioural therapy).

Recently, the application of Pain Neuroscience Education (PNE) as an intervention on its own, as well as in combination with another form of therapy (such as physiotherapy or cognitive- behavioural therapy) is receiving growing interest in the pediatric field of chronic pain. PNE aims to make people understand how their pain is produced and enables them to integrate this understanding into their everyday lives and subsequent treatment components. This innovative education style has shown to be effective in various adult chronic pain populations, by improving the patients' pain coping strategies and health status, and changing their pain beliefs. Although, no study examined the effectiveness of PNE in the context of chronic pediatric pain.

The hypothetical efficacy of pediatric PNE is based on previous findings in adult research that a better understanding of the nature of the illness results in improved patient outcomes. When children do not understand the origin of their pain, they might develop irrational beliefs and fears (including catastrophizing) about their pain, sustaining the vicious circle of chronic pain. Indeed, the information and context in which children perceive their pain, has been shown to modulate pain expectations and emotional response to pain. Since research findings showed that even parental beliefs about the aetiology of the child's pain influences the child's pain outcomes, the role of parents as 'pain modulators' might not be underestimated. Therefore, parents should be involved during PNE.

Concrete, the present study will examine whether reconceptualization of pain, by PNE is able to influence both child and parent knowledge of pain, as well as some other pain-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children
2. Informed consent

Exclusion Criteria:

1. Previous pain education
2. Chronic pain
3. Insufficient knowledge of the Dutch language
4. Mental retardation
5. Parent with chronic pain

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
Dutch Pediatric Neurophysiology of Pain Questionnaire (PedNPQ) | Change from baseline (before PNE) to immediately after PNE and 1 week following PNE
  The neurophysiology of pain knowledge of the child and parent will be assessed by using a questionnaire. The Dutch Pediatric Neurophysiology of Pain Questionnaire (PedNPQ) will be used to determine the current knowledge of pain and to evaluate the effect of PNE.
Neurophysiology of Pain Questionnaire (NPQ) | Change from baseline (before PNE) to immediately after PNE and 1 week following PNE
  The parent's knowledge of pain will also be assessed by the Neurophysiology of Pain Questionnaire (NPQ).

SECONDARY OUTCOMES:
Pain-related fear using the Fear of Pain Questionnaire - Parent version (FOPQ-P) | Baseline (before PNE) and 1 week following PNE
  For parental report, the Fear of Pain Questionnaire - Parent version (FOPQ-P) will be used to assess their own fear and avoidance behavior associated with their child's pain.
Catastrophic thinking about pain using the Dutch version of the Pain Catastrophizing Scale (PCS) | Baseline (Before PNE) and 1 week following PNE
  Catastrophic thinking about pain will be measured using the Dutch version of the Pain Catastrophizing Scale (PCS).
  Parent's catastrophic thinking about their child's pain will be measured using the Dutch version of the Pain Catastrophizing Scale for Parents (PCS-P).
Pain Vigilance and Awareness assessed by the Pain Vigilance and Awareness Questionnaire (PVAQ) | Baseline (before PNE) and 1 week following PNE
  Pain vigilance and awareness of the parent will be assessed by the Pain Vigilance and Awareness Questionnaire (PVAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Roselien Pas, MSc, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Pergolizzi J, Ahlbeck K, Aldington D, Alon E, Coluzzi F, Dahan A, Huygen F, Kocot-Kepska M, Mangas AC, Mavrocordatos P, Morlion B, Muller-Schwefe G, Nicolaou A, Perez Hernandez C, Sichere P, Schafer M, Varrassi G. The development of chronic pain: physiological CHANGE necessitates a multidisciplinary approach to treatment. Curr Med Res Opin. 2013 Sep;29(9):1127-35. doi: 10.1185/03007995.2013.810615. Epub 2013 Jul 3. PMID 23786498
- [Background] Goodman JE, McGrath PJ. The epidemiology of pain in children and adolescents: a review. Pain. 1991 Sep;46(3):247-264. doi: 10.1016/0304-3959(91)90108-A. No abstract available. PMID 1758709
- [Background] Simons LE, Basch MC. State of the art in biobehavioral approaches to the management of chronic pain in childhood. Pain Manag. 2016;6(1):49-61. doi: 10.2217/pmt.15.59. Epub 2015 Dec 17. PMID 26678858
- [Background] Korterink JJ, Diederen K, Benninga MA, Tabbers MM. Epidemiology of pediatric functional abdominal pain disorders: a meta-analysis. PLoS One. 2015 May 20;10(5):e0126982. doi: 10.1371/journal.pone.0126982. eCollection 2015. PMID 25992621
- [Background] Roth-Isigkeit A, Thyen U, Stoven H, Schwarzenberger J, Schmucker P. Pain among children and adolescents: restrictions in daily living and triggering factors. Pediatrics. 2005 Feb;115(2):e152-62. doi: 10.1542/peds.2004-0682. PMID 15687423
- [Background] Vervoort T, Logan DE, Goubert L, De Clercq B, Hublet A. Severity of pediatric pain in relation to school-related functioning and teacher support: an epidemiological study among school-aged children and adolescents. Pain. 2014 Jun;155(6):1118-1127. doi: 10.1016/j.pain.2014.02.021. Epub 2014 Mar 12. PMID 24631587
- [Background] Landry BW, Fischer PR, Driscoll SW, Koch KM, Harbeck-Weber C, Mack KJ, Wilder RT, Bauer BA, Brandenburg JE. Managing Chronic Pain in Children and Adolescents: A Clinical Review. PM R. 2015 Nov;7(11 Suppl):S295-S315. doi: 10.1016/j.pmrj.2015.09.006. PMID 26568508
- [Background] Goddard JM. Chronic pain in children and young people. Curr Opin Support Palliat Care. 2011 Jun;5(2):158-63. doi: 10.1097/SPC.0b013e328345832d. PMID 21415756
- [Background] Robins H, Perron V, Heathcote LC, Simons LE. Pain Neuroscience Education: State of the Art and Application in Pediatrics. Children (Basel). 2016 Dec 21;3(4):43. doi: 10.3390/children3040043. PMID 28009822
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Van Oosterwijck J, Meeus M, Paul L, De Schryver M, Pascal A, Lambrecht L, Nijs J. Pain physiology education improves health status and endogenous pain inhibition in fibromyalgia: a double-blind randomized controlled trial. Clin J Pain. 2013 Oct;29(10):873-82. doi: 10.1097/AJP.0b013e31827c7a7d. PMID 23370076
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Meeus M, Nijs J, Van Oosterwijck J, Van Alsenoy V, Truijen S. Pain physiology education improves pain beliefs in patients with chronic fatigue syndrome compared with pacing and self-management education: a double-blind randomized controlled trial. Arch Phys Med Rehabil. 2010 Aug;91(8):1153-9. doi: 10.1016/j.apmr.2010.04.020. PMID 20684894
- [Background] Jackson T, Pope L, Nagasaka T, Fritch A, Iezzi T, Chen H. The impact of threatening information about pain on coping and pain tolerance. Br J Health Psychol. 2005 Sep;10(Pt 3):441-51. doi: 10.1348/135910705X27587. PMID 16238858
- [Background] Boerner KE, Noel M, Birnie KA, Caes L, Petter M, Chambers CT. Impact of Threat Level, Task Instruction, and Individual Characteristics on Cold Pressor Pain and Fear among Children and Their Parents. Pain Pract. 2016 Jul;16(6):657-68. doi: 10.1111/papr.12306. Epub 2015 May 26. PMID 26011606
- [Background] Palermo TM, Chambers CT. Parent and family factors in pediatric chronic pain and disability: an integrative approach. Pain. 2005 Dec 15;119(1-3):1-4. doi: 10.1016/j.pain.2005.10.027. Epub 2005 Nov 18. No abstract available. PMID 16298492